CLINICAL TRIAL: NCT06912321
Title: Construction of Papez Loop Neural Network Feature Recognition Model and Prediction Model of Cognitive Impairment Progression Related to Insulin Resistance in Type 2 Diabetes Mellitus
Brief Title: Characteristics of Papez Loop Neural Network in T2DM （Type 2 Diabetes Mellitus）
Acronym: T2DM
Status: Recruiting | Type: Observational
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: KY20240419-04-KS-01
Record Dates: First submitted 2024-05-23; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-02

CONDITIONS: Type 2 Diabetes; Insulin Resistance; Cognitive Impairment
Keywords: Type 2 Diabetes; Insulin Resistance; Papez circuit; Multimodal magnetic resonance imaging; Machine learning
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Type 2 Diabetes: These patients must have a definite diagnosis of type 2 diabetes mellitus (T2DM) according to the American Diabetes Association (ADA) standards
  Interventions: Other: No Intervention: Observational Cohort
- Healthy control: These participants have normal glucose tolerance and normal cognition
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No Intervention: Observational Cohort — No intervention：all participants did not receive any intervention measures throughout the study

SUMMARY:
This is a cross-sectional and longitudinal study to investigate the characteristic changes in Papez's circuit neural network activity and connectivity based on multimodal MRI, and through follow-up study of the interaction between the internal brain regions of Papez circuit and the function of the external neural network, a prediction model of the characteristic changes of Papez circuit neural network was constructed based on machine learning technology.

DETAILED DESCRIPTION:
T2DM patients may have multidimensional cognitive impairment, which is related to the damage of key brain regions in Papez's circuit. The purpose of this study is to establish a prediction model for the occurrence, development, and severity of cognitive impairment by using machine learning of Papez circuit neural network in T2DM patients. This will allow for early intelligent assessment with high accuracy and efficiency, and assist in clinical personalized treatment and early intervention. The research center has 1 principal investigator, 4 sub-investigators, and 1 nurse. Participants will include 200 patients with type 2 diabetes recruited from outpatient and inpatient departments. Additionally, 200 healthy controls will be recruited from the community. Each subject will undergo clinical information collection, biochemical measurements including fasting blood glucose, C-peptide, HbA1c, blood lipid, postprandial blood glucose, and postprandial C-peptide, multimodal MRI scans, and cognitive assessments at baseline and each follow-up visit. The study duration is 6 years, with a follow-up every 36 months. At the end of the study, all assessments will be performed again for all recruited subjects.

ELIGIBILITY:
Inclusion Criteria:

1. T2DM patients met the diagnostic criteria for diabetes (WHO, 1999) with a duration of 3-20 years; The control group met the criteria of fasting blood glucose < 6.1mmol/l and glycosylated hemoglobin < 5.7%;
2. right-handed, aged 45-70 years, with ≥8 years of education;
3. no contraindications to MRI scanning such as electronic and metal device implantation;
4. The visual acuity or corrected visual acuity and binaural hearing can meet the needs of the evaluation, and can cooperate to complete the examination.
5. without a history of substance abuse or dependence, evaluation is not used during the period of calm sleeping pills and antidepressants, not long-term use of drugs to improve cognitive.

Exclusion Criteria:

1. patients with acute metabolic complications or a history of severe hypoglycemia;
2. severe heart, liver, lung, kidney and hematopoietic system diseases; Hyperthyroidism or hypothyroidism; Stroke, alzheimer's disease, epilepsy, Parkinson's disease and other neurological history; A history of mental illness such as depression, mania, or alcohol dependence; History of loss of consciousness due to neurological diseases or traumatic brain injury;
3. one month before the laboratory examination, with a record and surgical trauma infection;

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: T2DM patients will be recruited from the outpatient and inpatient units of the endocrinology department of the investigator's hospital. Healthy control will be recruited in the community
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2030-05-01 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Baseline brain structural MRI scan | Within 1 week after neuropsychological tests
  To calculate the volumes of whole brain and target brain regions
Baseline brain functional MRI scan | Within 1 week after neuropsychological tests
  To evaluate Papez loop cross-scale network variation
Baseline brain diffusion tensor MRI scan | Within 1 week after neuropsychological tests
  To trace and reconstruct the nerve fiber tracts between the Papez circuit related brain regions and between the circuit and the outer brain regions, and to construct a structural connection network according to the characteristics of white matter conduction pathways
Baseline brain arterial spin labeling MRI scan | Within 1 week after neuropsychological tests
  To calculate the blood perfusion in the whole brain and Papez circuit
Baseline neuropsychological performance | Day 1 of entry study
  Montreal Cognitive Assessment，MoCA：It includes 11 examination items in 8 cognitive domains with a total score of 30 points
Baseline neuropsychological performance | Day 1 of entry study
  Mini-mental State Examination，MMSE：The highest score is 30 points, with scores between 27-30 indicating normal and scores below 27 indicating cognitive impairment
Baseline neuropsychological performance | Day 1 of entry study
  Complex Figure Test, CFT: The total score is 36 points, including position score and shape score
Baseline neuropsychological performance | Day 1 of entry study
  Verbalfluencytest, VFT: includes semantic fluency test, speech fluency test, and action fluency test
Baseline neuropsychological performance | Day 1 of entry study
  Trail making testTMT：includes two parts, A and B
Baseline neuropsychological performance | Day 1 of entry study
  Auditory Verbal Learning Test， VALT
Baseline neuropsychological performance | Day 1 of entry study
  Digit span test,DST
Baseline neuropsychological performance | Day 1 of entry study
  Digit Symbol Substitution Test, DSST
Baseline peripheral blood neuropathology biomarkers level | Blood samples will be collected on day 1 of the entry study
  Fasting blood glucose（mmol/L）
Baseline peripheral blood neuropathology biomarkers level | Blood samples will be collected on day 1 of the entry study
  C-peptide（nmol/l）
Baseline peripheral blood neuropathology biomarkers level | Blood samples will be collected on day 1 of the entry study
  HbA1c（mmol/mol）
Baseline peripheral blood neuropathology biomarkers level | Blood samples will be collected on day 1 of the entry study
  blood lipid（mmol/L）
Baseline peripheral blood neuropathology biomarkers level | Blood samples will be collected on day 1 of the entry study
  postprandial blood glucose（mmol/L）
Baseline peripheral blood neuropathology biomarkers level | Blood samples will be collected on day 1 of the entry study
  postprandial C-peptide（nmol/l）

SECONDARY OUTCOMES:
Longitudinal changes of brain structural MRI scan | 36 months, 72 months
  Compare the changes of the volumes of whole brain and target brain regions from baseline to each follow-up time points
Longitudinal changes of brain functional MRI scan | 36 months, 72 months
  Compare the changes of the Papez circuit cross-scale network variation from baseline to each follow-up time points
Longitudinal changes of brain diffusion tensor MRI scan | 36 months, 72 months
  Compare the changes of the Papez circuit structural network from baseline to each follow-up time points
Longitudinal changes of brain arterial spin labeling MRI scan | 36 months, 72 months
  Compare the changes of blood perfusion in the whole brain and Papez circuit from baseline to each follow-up time points
Longitudinal changes of neuropsychological performance | 36 months, 72 months
  Compare the Montreal Cognitive Assessment(MoCA) change from the baseline to each follow-up time points
Longitudinal changes of neuropsychological performance | 36 months, 72 months
  Compare the Mini-mental State Examination (MMSE) change from the baseline to each follow-up time points
Longitudinal changes of neuropsychological performance | 36 months, 72 months
  Compare the Complex Figure Test (CFT) change from the baseline to each follow-up time points
Longitudinal changes of neuropsychological performance | 36 months, 72 months
  Compare the Verbalfluencytest (VFT) change from the baseline to each follow-up time points
Longitudinal changes of neuropsychological performance | 36 months, 72 months
  Compare the Trail making test (TMT) change from the baseline to each follow-up time points; includes two parts, A and B
Longitudinal changes of neuropsychological performance | 36 months, 72 months
  Compare the Auditory Verbal Learning Test (VALT) change from the baseline to each follow-up time points
Longitudinal changes of neuropsychological performance | 36 months, 72 months
  Compare the Digit span test (DST) change from the baseline to each follow-up time points
Longitudinal changes of neuropsychological performance | 36 months, 72 months
  Compare the Digit Symbol Substitution Test (DSST) change from the baseline to each follow-up time points
Longitudinal changes of peripheral blood neuropathology biomarkers leve | 36 months, 72 months
  Compare the fasting blood glucose（mmol/L）changes from baseline to each follow-up time points
Longitudinal changes of peripheral blood neuropathology biomarkers leve | 36 months, 72 months
  Compare the C-peptide（nmol/l）changes from baseline to each follow-up time points
Longitudinal changes of peripheral blood neuropathology biomarkers leve | 36 months, 72 months
  Compare the HbA1c（mmol/mol）changes from baseline to each follow-up time points
Longitudinal changes of peripheral blood neuropathology biomarkers leve | 36 months, 72 months
  Compare the blood lipid（mmol/L）changes from baseline to each follow-up time points
Longitudinal changes of peripheral blood neuropathology biomarkers leve | 36 months, 72 months
  Compare the postprandial blood glucose（mmol/L）changes from baseline to each follow-up time points
Longitudinal changes of peripheral blood neuropathology biomarkers leve | 36 months, 72 months
  Compare the postprandial C-peptide（nmol/l）changes from baseline to each follow-up time points
Machine learning of multimodal MRI data | 72 months
  Multimodal MRI data for machine learning, can be in different levels of calculation and analysis and research on the characteristics of neural network, found a pattern classification and predict unknown data effectively, find out the Papez loop associated with insulin resistance characteristics of neural network

CONTACTS AND LOCATIONS:
Overall Officials: Wenqing Xia, PHD, Study Chair — Department of Endocrinology, Nanjing First Hospital, Nanjing Medical University, Nanjing, China
Locations (1):
- Department of Endocrinology, Nanjing First Hospital, Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided